CLINICAL TRIAL: NCT01885364
Title: Esmolol Pretreatment on Pain During Injection of Propofol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kyungpook National University Hospital (Other)
Responsible Party: Principal Investigator, Younghoon Jeon, Associate Professor, Kyungpook National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: KNUH 2013-05-003-001
Record Dates: First submitted 2013-06-18; First posted 2013-06-25 (Estimated); Last update posted 2016-02-08 (Estimated); Status verified 2016-02

CONDITIONS: Pain
Keywords: esmolol; pain; propofol; remifentanil
MeSH Terms: conditions — Pain | interventions — Saline Solution; esmolol; Remifentanil; Propofol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Placebo & propofol (Placebo Comparator): Pretreatment with normal saline before injection of propofol
  Interventions: Drug: Normal saline; Drug: propofol
- esmolol 0.05 mg/kg & propofol (Experimental): Pretreatment with esmolol 0.05 mg/kg before injection of propofol
  Interventions: Drug: Esmolol; Drug: propofol
- esmolol 1 mg/kg & propofol (Experimental): Pretreatment with esmolol 1 mg/kg before injection of propofol
  Interventions: Drug: Esmolol; Drug: propofol
- remifentanil 0.35 ug/kg & propofol (Active Comparator): Pretreatment with remifentanil 0.35 ug/kg before injection of propofol
  Interventions: Drug: Remifentanil; Drug: propofol

INTERVENTIONS:
Drug: Normal saline — intravenous injection with normal saline before injection of propofol
  Arms: Placebo & propofol
Drug: Esmolol — intravenous injection with remifentanil 0.5 mg/kg before injection of propofol
  Other Names: breviblock
  Arms: esmolol 0.05 mg/kg & propofol; esmolol 1 mg/kg & propofol
Drug: Remifentanil — intravenous injection with remifentanil 0.35 ug/kg before injection of propofol
  Other Names: ultiva
  Arms: remifentanil 0.35 ug/kg & propofol
Drug: propofol — intravenous injection after pretreatment
  Other Names: diprivan

SUMMARY:
Pain on injection of propofol is a common side effect. The present study was designed to investigate the effect of esmolol on pain on propofol injection and to compare it with remifentanil and placebo.

DETAILED DESCRIPTION:
In a double-blind, prospective trial, 120 patients scheduled to undergo elective surgery were randomized to receive normal saline (n=30), remifentanil 0.35 μg/kg (n=30), esmolol 0.5 mg/kg (n=30), or Esmolol 1mg/kg (n=30) as pretreatment. Thirty seconds after pretreatment, 25% of the total calculated dose of propofol (2 mg/kg) was administrated into a dorsal hand vein. Ten seconds after propofol had been given at the rate of 0.5 ml/sec pain was assessed on a four-point scale (0=none, 1 = mild, 2= moderate, 3= severe).

ELIGIBILITY:
Inclusion Criteria:

* patients aged 19-60 years, American Society of Anesthesiologists (ASA) physical status I and II, scheduled for elective surgery under general anesthesia

Exclusion Criteria:

* Patients with cardiovascular, neurological or psychiatric disorder problem, patients who received the analgesic or sedative medications within the last 24 hours, and pregnancy were excluded

Ages: 19 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2015-06; Primary Completion 2015-11 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Pain on injection of propofol | 10 seconds after injection of 25% of the total calculated dose of propofol (2 mg/kg)
  Thirty seconds after pretreatment, 25% of the total calculated dose of propofol (2 mg/kg) was administrated into a dorsal hand vein. Ten seconds after injection of propofol, pain was assessed on a four-point scale (0=none, 1 = mild, 2= moderate, 3= severe).

CONTACTS AND LOCATIONS:
Overall Officials: Younghoon Jeon, Dr, Principal Investigator — Kyungpook National University Hospital
Locations (1):
- Kyungpook National University Hospital, Daegu, South Korea